CLINICAL TRIAL: NCT03750656
Title: Use of Hyoscyamine Versus Tamsulosin for Management of Ureteral Stent Irritation
Acronym: HyTa Stent
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not accruing patients quickly enough
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, David Duchene, MD, Associate Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC 142994
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Lower Urinary Tract Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Hyoscyamine; Tamsulosin

STUDY DESIGN:
Intervention Model Description: Randomized open-blind clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyoscyamine (Active Comparator): Hyoscyamine 0.125 mg tab sublingual every 4 hours as needed for discomfort
  Interventions: Drug: Hyoscyamine
- Tamsulosin (Active Comparator): 0.4 mg tab orally daily
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Hyoscyamine — Patients will be randomized to receive hyoscyamine for lower urinary tract symptoms are placement of ureteral stent
  Arms: Hyoscyamine
Drug: Tamsulosin — Patients will be randomized to receive tamsulosin for lower urinary tract symptoms are placement of ureteral stent
  Arms: Tamsulosin

SUMMARY:
The objective of this project is to compare the efficacy of hyoscyamine to tamsulosin monotherapy in treating lower urinary tract symptoms in patients with indwelling double-J ureteral stents.

DETAILED DESCRIPTION:
Ureteral stents are routinely used in a variety of urologic conditions. Unfortunately, indwelling ureteral stents commonly cause significant pain and discomfort due to irritation to the urinary system. Many studies have looked at methods to reduce these uncomfortable symptoms ranging from altering stent designs to pharmacologic therapies attempting to alleviate stent-discomfort. However, stent-related discomfort continues to be an issue and is often the cause of their removal earlier than planned. While the efficacy of certain alpha blockers and anticholinergics in treating stent-related symptoms have been studied, the data for the use of hyoscyamine in this setting is lacking. A literature search yielded no studies evaluating the use of hyoscyamine in this setting to date. The investigators hypothesize that hyoscyamine (brand name Levsin) is equivalent to tamsulosin in treating lower urinary tract symptoms in patients with indwelling double-J ureteral stents due to its anticholinergic properties. Furthermore, the investigators hypothesize that patients in the hyoscyamine arm will not require additional pain medications (e.g. Pyridium, narcotics) to help control stent-related discomfort compared to the tamsulosin arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Patient must require placement of a ureteral stent(s), per standard of care, following routine urological procedures including, but not limited to, ureteroscopy, stone extraction, or management of upper tract transitional cell carcinoma
* Patient must agree to abstain from other clinical studies during the study period

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients with chronic or pre-existing indwelling stents
* Patients currently receiving anticholinergic or alpha blocker therapy
* Patients with chronic opioid or analgesic usage
* Patients with chronic pain syndrome or symptomatic benign prostatic hyperplasia
* Patients with an active untreated urinary tract infection
* Patients who are currently pregnant or nursing
* Patients with allergies or contraindication to either tamsulosin or hyoscyamine
* Patients on active chemotherapy
* Patients currently receiving other investigational therapy
* Patients who are unable to sign consent/answer questionnaire due to compromised mental capacity or language barrier (the questionnaire is not validated in other languages)
* Patients who have a stent placed emergently for an obstructing stone or septic stone without immediate stone removal,
* Any stents placed that will stay in for longer than 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyoscyamine | Tamsulosin
Started | 4 | 1
Completed | 2 | 0
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyoscyamine | Tamsulosin | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Ureteral Stent Symptom Questionnaire Score
Description: To evaluate the efficacy of hyoscyamine compared to tamsulosin in improving the lower urinary tract symptoms of patients with indwelling double-J ureteral stents as assessed by the validated Ureteral Stent Symptom Questionnaire (USSQ).
Time Frame: Three Years
Population: Data not collected to complete data analysis for the patients enrolled.
Arm/Group | Hyoscyamine | Tamsulosin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Additional Medication Needed
Description: To determine if there is a difference between the amount of additional medications needed to treat stent related discomfort between patients receiving hyoscyamine versus those that receive tamsulosin
Time Frame: Three Years
Population: Data not collected to complete data analysis for the patients enrolled.
Arm/Group | Hyoscyamine | Tamsulosin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Factors That Determine if Additional Medication Needed
Description: To determine factors contributing to patients needing additional medication for treatment of stent-related discomfort
Time Frame: Three Years
Population: Data not collected to complete data analysis for the patients enrolled.
Arm/Group | Hyoscyamine | Tamsulosin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Not Applicable - Adverse events were not documented.
Description: Study was terminated early therefore no data was collected to monitor/assess adverse events.
Arm/Group | Hyoscyamine | Tamsulosin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03750656/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT03750656/ICF_001.pdf